CLINICAL TRIAL: NCT05183568
Title: Mindful Self-Compassion (MSC) as an Intervention for Infertility Related Distress: A Pilot Study
Brief Title: Mindful Self-Compassion (MSC) for Infertility Related Distress
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Principal Investigator, Jennifer Gordon, Associate professor, University of Regina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB #2021-133
Record Dates: First submitted 2021-12-07; First posted 2022-01-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2021-12

CONDITIONS: Infertility, Female; Distress, Emotional; Depressive Symptoms; Anxiety
MeSH Terms: conditions — Infertility, Female; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mindful Self-Compassion (Experimental): Participants will undergo an 8-week self-help program consisting of assigned weekly chapters in the workbook entitled "The Mindful Self-Compassion Workbook: A Proven Way to Accept Yourself, Build Inner Strength, and Thrive" (Neff & Germer, 2018), paired with daily guided meditations provided through a free smartphone app that was developed by the Centre for Mindfulness Studies, a Canadian-based mental health charity.
  Interventions: Behavioral: Mindful Self-Compassion

INTERVENTIONS:
Behavioral: Mindful Self-Compassion — Self-guided bibliotherapy (specific chapters to read each week) and daily use of a meditation app for 45 minutes

SUMMARY:
This study will test a psychological intervention for the treatment of distress related to infertility. The intervention will pair reading a book "The Mindful Self-Compassion Workbook" by Kristin Neff with guided meditations using the Centre for Mindfulness Studies mobile app. Individuals with infertility will complete the 8-week program and complete psychological outcome measures before and after.

DETAILED DESCRIPTION:
The investigators will recruit 50 women struggling with infertility across Canada and the United States via a paid Facebook ad as well as advertising via online infertility support groups. Participants will undergo an 8-week self-help program consisting of assigned weekly chapters in the workbook entitled "The Mindful Self-Compassion Workbook: A Proven Way to Accept Yourself, Build Inner Strength, and Thrive" (Neff & Germer, 2018), paired with daily guided meditations provided through a free smartphone app that was developed by the Centre for Mindfulness Studies, a Canadian-based mental health charity. The app is free to download on the app store for iPhone and Android. After completing a Zoom-faciliated enrollment session during which eligibility will be confirmed and informed consent obtained, participants will be mailed a copy of the workbook and instructed to complete three chapters per week for a total eight weeks. Each chapter is approximately 5-7 pages long but includes reflection exercises that may take some time - each chapter is therefore expected to take participants approximately 20 minutes to read. Participants will be sent a weekly email to remind them of their assigned chapters to read each week by the graduate student researcher.

Before starting the program, participants will be asked to complete a demographics form and the Credibility/Expectancy Questionnaire (CEQ) pre-intervention, as well as a series of questionnaires both before and after the intervention. The questionnaires are as follows: Fertility Quality of life Questionnaire (FertQoL), State-Trait Anxiety Inventory (STAI), the Generalised Anxiety Disorder-7 (GAD-7), Patient Health Questionnaire-9 (PHQ-9), The Five Facet Mindfulness Questionnaire-15 (FFMQ-15), The Self-Compassion Scale, The Compassion Scale, the Revised Dyadic Adjustment Scale (RDAS) and a brief survey about what participants liked or disliked about the program. These surveys will be completed at baseline, at the end of the 8th intervention week, and then one month after the program is over. Participants' app usage will be tracked by the Centre for Mindfulness Studies and shared with our research team, allowing us to assess adherence to the assigned homework.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Undergoing fertility treatments or who have failed to conceive despite a 12 month period without the use of contraception
* Reporting distress related to infertility, as indicated by Fertility Quality of Life Questionnaire score below 70, which is indicative of below-average quality of life

Exclusion Criteria:

* Currently seeking psychological treatment
* Participation in a formal mindfulness program within 6 months of recruitment
* Endorsement of active suicidal ideation, indicated by a score of 8 or above on the Suicidal Behaviors Questionnaire
* GAD-7 score of 15-21, indicating severe generalized anxiety
* PHQ-9 score of 20-27, indicating severe depressive symptoms.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Fertility-related quality of life | Immediately post-intervention
  Score on the FertiQoL (fertility-related Quality of Life tool) - scores range from 0 to 100 and higher scores indicate better quality of life
Fertility-related quality of life | 1 month post-intervention
  Score on the FertiQoL (fertility-related Quality of Life tool) - scores range from 0 to 100 and higher scores indicate better quality of life

SECONDARY OUTCOMES:
Anxious symptoms | Immediately post-intervention
  Scores on the GAD-7 (Generalized Anxiety Disorder-7) - scores range from 0 to 21 and higher scores indicate more severe anxiety
Anxious symptoms | 1 month post-intervention
  Scores on the GAD-7 (Generalized Anxiety Disorder-7) - scores range from 0 to 21 and higher scores indicate more severe anxiety
Depressive symptoms | Immediately post-intervention
  Scores on the PHQ-9 (Patient History Questionnaire-9) - scores range from 0 to 27 and higher scores indicate more severe symptoms
Depressive symptoms | 1 month post-intervention
  Scores on the PHQ-9 (Patient History Questionnaire-9) - scores range from 0 to 27 and higher scores indicate more severe symptoms

OTHER OUTCOMES:
Trait mindfulness | Immediately post-intervention
  Scores on the FFMQ-15 (Five Facet Mindfulness Questionnaire-15) - scores range from 3 to 15 and higher scores indicate higher levels of mindfulness
Trait mindfulness | 1 month post-intervention
  Scores on the FFMQ-15 (Five Facet Mindfulness Questionnaire-15) - scores range from 3 to 15 and higher scores indicate higher levels of mindfulness
Trait self-compassion | Immediately post-intervention
  Scores on the SCS (Self-Compassion Scale) - scores range from 1 to 5, with higher scores indicating higher self-compassion
Trait self-compassion | 1 month post-intervention
  Scores on the SCS (Self-Compassion Scale) - scores range from 1 to 5, with higher scores indicating higher self-compassion
Relationship quality | Immediately post-intervention
  Scores on the RDAS (Revised Dyadic Adjustment Scale) - scores range from 0 to 69 and higher scores indicate better relationship quality
Relationship quality | 1 month post-intervention
  Scores on the RDAS (Revised Dyadic Adjustment Scale) - scores range from 0 to 69 and higher scores indicate better relationship quality

CONTACTS AND LOCATIONS:
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No